CLINICAL TRIAL: NCT00462241
Title: Non-cardiac Chest Pain Evaluation and Treatment Study (CARPA) - Part 2: Treatment Study
Brief Title: Treatment Study Comparing Manual Treatment or Advice in Acute, Musculoskeletal Chest Pain
Acronym: CARPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Locomotion Science (Other)
Collaborators: Nordic Institute of Chiropractic and Clinical Biomechanics (Other); Odense University Hospital (Other); University of Southern Denmark (Other); The County of Funen, Denmark (Other Government); Foundation for Chiropractic Research and Post Graduate Education (Other)
Responsible Party: Principal Investigator, Mette Jensen Stochkendahl, DC, PhD, Clinical Locomotion Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project 73 - RCT (NMA)
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Musculoskeletal Chest Pain; Non-cardiac Chest Pain; Undiagnosed Chest Pain
Keywords: Chest pain; Chest wall; Atypical chest pain; Non-cardiac chest pain; Undiagnosed chest pain; Physical examination; Randomized controlled trial; Treatment study; Chiropractor
MeSH Terms: conditions — Chest Pain | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chiropractic treatment (Experimental): Individualised chiropractic treatment, pragmatic approach
  Interventions: Procedure: chiropractic treatment
- self-management (Sham Comparator): Self-management: Minimal intervention - practice as usual.
  Interventions: Other: Self-management

INTERVENTIONS:
Procedure: chiropractic treatment — Participants in the therapy group undergo a physical examination by an experienced, primary sector chiropractor, lasting up to one hour. The chiropractors choose an individual treatment strategy based on a combination of their findings, the patient history, and a standardized protocol reflecting routine practice. The standardized treatment protocol includes high velocity, low amplitude manipulation directed towards the thoracic and/or cervical spine in combination with any of the following: Joint mobilisation, soft tissue techniques, stretching, stabilising or strengthening exercises, heat or cold treatment, and advice. The protocol specifies up to ten treatment sessions of approximately 20 minutes, 1-3 times per week, or treatment until the patient is pain free. The chiropractors record the types of treatment rendered at sessions.
  Arms: chiropractic treatment
Other: Self-management — Advice group: Advice is directed towards promoting self-management. The participants are told that their chest pain generally has a benign, self limiting course. The participants receive individual instructions regarding posture and two or three exercises aiming to increase spinal or muscle stretch based on clinical evaluation. They are advised to seek medical attention for re-evaluation (general physician, chest pain clinic or emergency department) in case of severe or unfamiliar chest pain. The session lasts on average 15 minutes. Further, the advice group is also asked not to seek any manual treatment for the next four weeks.
  Arms: self-management

SUMMARY:
Acute chest pain is a common cause of hospital admission. Active approaches are directed towards diagnosis and treatment of potentially life threatening conditions, especially acute coronary syndrome and coronary artery disease. However, a considerable number of patients may have chest pain caused by biomechanical dysfunction of muscles and joints of the chest wall or the cervical and thoracic spine (20%). The diagnostic approaches and treatment options for this group of patients are scarce and there is a lack of formal clinical studies and validated outcome measures addressing the effect of manual treatment approaches.

Objective: This single blind randomized clinical trial investigates whether chiropractic treatment can reduce pain and improve function in a population of patients with acute, musculoskeletal chest pain when compared to advice directed towards promoting self-management.

Methods: Among patients admitted to a chest pain clinic in a university hospital under suspicion of acute coronary syndrome, 120 patients with an episode of acute chest pain of musculoskeletal origin are included in the study. All patients have completed the chest pain clinic diagnostic procedures, and acute coronary syndrome and other obvious reasons for chest pain have been excluded. After completion of the study evaluation program, the patients are randomized into one of two groups: A) advice promoting self-management and individual instructions focusing on posture and muscle stretch; B) a course of chiropractic therapy of up to ten treatment sessions focusing on high velocity, low amplitude manipulation of the cervical and thoracic spine together with a choice of mobilisation and soft tissue techniques. In order to establish suitable outcome measures, two pilot studies were conducted. Outcome measures are pain, function, overall health, and patient-rated treatment effect measured at 4, 12, and 52 weeks following treatment.

DETAILED DESCRIPTION:
BACKGROUND

Acute chest pain is one of the most common reasons for hospital admission.(Bechgaard, 1982) In Denmark alone, more than 30,000 patients are admitted to medical departments because of chest pain.(Fruergaard, 1992) In the United States chest pain is the reason for 20-30 percent of all acute medical hospital admissions.(Capewell, 2000) However, an estimated 5-20 percent of all admissions to acute chest pain departments are caused by chest pain of musculoskeletal origin.(Knockaert 2002; Spalding 2003; Fruergaard 1996)

Chest pain patients with normal coronary anatomy have an excellent prognosis for survival and a future risk of cardiac morbidity similar to that reported in the background population.(Berman 1999; Klocke 2003) However, about three quarters of patients with non-cardiac chest pain continue to suffer from residual chest pain with large socio-economic consequences.(Spalding 2003; Launbjerg 1997; Ockene 1980; Eslick 2002; Tew 1995; Wielgosz 1984; Achem 2000)

An extensive body of literature addresses patient management protocols for patients presenting with chest pain primarily focusing on cardiopulmonary, gastroesophageal, and psychological conditions causing chest symptoms, but treatment protocols of musculoskeletal chest pain remain, however, scarce. Neither the effect of medical treatment (oral anti-inflammatory drug), exercise (strength and/or stretching), nor advice have been investigated. In particular, there is a lack of formal clinical studies examining the effectiveness of manual/manipulative approaches to manage musculoskeletal chest pain. To the best of the authors knowledge, only one study exists that deal with this aspect.(Christensen, 2005)

Therefore, the aim of this single-blind randomized clinical trial is to compare the effect of chiropractic treatment versus advice directed towards promoting self-management in a population of patients with musculoskeletal chest pain using standardized outcome measures. Further, a cost-effectiveness analysis along side the RCT will be performed.

METHODS

Design: Single-blinded Randomized Trial.

Study sample:

The patients are recruited from a university hospital chest pain clinic. The chest pain clinic is part of a large specialized cardiology department. All patients undergo a standardized evaluation program ruling out acute coronary syndrome and any other obvious and significant cardiac or non-cardiac disease. Sixty patients are to be included in each of the two intervention groups, totaling 120 participants. The patients are included as a part of a larger study on diagnosis of musculoskeletal chest pain.

Examination and baseline data:

Following discharge from the chest pain clinic, all patient records are screened for the inclusion and non-inclusion criteria, and potential participants are invited to participate. Within 7 days, participants are assessed in an individual baseline test. First, they complete a battery of questionnaires including information on social, occupation, education, physical and lifestyle factors, expectation to treatment outcome, and baseline values for the outcome measure (see below). Signed consent forms are obtained from all participants.

Next, patients with musculoskeletal chest pain will be identified using a standardized examination protocol. The examination protocol consists of 3 parts: 1) a semi-structured interview (including pain characteristics, symptoms from the lungs and gastrointestinal system, the past medical history, height and weight, and risk factors of ischemic heart disease), 2) a general health examination (including blood pressure and pulse, heart and lung stethoscopy, abdominal palpation, neck auscultation, and clinical signs of left ventricular failure, neurological examination of upper and lower extremities in terms of reflexes, sensibility to touch, muscle strength, as well as orthopaedic examination of the neck and shoulder joints in order to rule out nerve root compression syndromes.), and 3) a specific manual examination of the muscles and joints of the neck, thoracic spine and thorax (including active range of motion, manual palpation for muscular tenderness on 14 point of the anterior chest wall, palpation for paraspinal muscular tenderness segmentally, motion palpation for joint-play restriction of the thoracic spine (Th1-8), and end play restriction of the cervical and thoracic spine).

The examination program together with the detailed case history will be applied by the clinician to the population of chest pain patients to make a diagnosis of pain from the musculoskeletal system, Cervico-thoracic Angina (CTA).

Randomization:

Only CTA positive participants draw a sealed, opaque envelope numbered in succession and containing information about treatment allocation. The randomization sequence is computer generated. The envelopes are arranged in clusters of varying size. The examining clinician manages the hand over of the envelope to the participant, but is blind to treatment allocation.

Interventions:

CTA positive participants will be randomized to receive advice promoting self-management (advice group) or a standard course of chiropractic treatment (therapy group).

Advice group: Advice is directed towards promoting self-management. The participants are told that their chest pain generally has a benign, self limiting course. The participants receive individual instructions regarding posture and two or three exercises aiming to increase spinal or muscle stretch based on clinical evaluation. They are advised to seek medical attention for re-evaluation (general physician, chest pain clinic or emergency department) in case of severe or unfamiliar chest pain. The session lasts on average 15 minutes. Further, the advice group is also asked not to seek any manual treatment for the next four weeks.

Therapy group: Participants in the therapy group undergo a physical examination by an experienced, primary sector chiropractor, lasting up to one hour. The chiropractors choose an individual treatment strategy based on a combination of their findings, the patient history, and a standardized protocol reflecting routine practice. The standardized treatment protocol includes high velocity, low amplitude manipulation directed towards the thoracic and/or cervical spine in combination with any of the following: Joint mobilization, soft tissue techniques, stretching, stabilizing or strengthening exercises, heat or cold treatment, and advice. The protocol specifies up to ten treatment sessions of approximately 20 minutes, 1-3 times per week, or treatment until the patient is pain free. The chiropractors record the types of treatment rendered at sessions.

Follow-up: Follow-up data are collected at four weeks, 3 months and one year (Figure 1)

Data analyzes: Data will be analyzed by a research group member blinded to group status. The analysis will be based on the intention to treat principle. Both parametric and non parametric principle will be used to compare treatment effects between the groups and to identify baseline predictors for successful treatment outcome. Finally, based on a prior definition of success, numbers needed to treat will be calculated.

Cost-effectiveness analysis: A cost comparison of the therapy and advice group will be performed using data on direct and indirect costs. A cost-utility analysis comparing the therapy and advice group will be performed using the EuroQol 5D.

ELIGIBILITY:
Inclusion Criteria:

To be included in the project the participant must

* Have chest pain as their primary complaint.
* Have an acute episode of pain of less than 7 days duration before admission.
* Consent to the standardized evaluation program at the chest pain clinic.
* Have pain the in the thorax and/or neck.
* Be able to read and understand Danish. Be between 18 and 75 year of age.
* Be a resident of the Funen County.

Patients will not be included if any of the following conditions are present

* ACS.
* Have had Percutaneous Coronary Intervention (PCI) or Coronary Artery By-pass Grafting (CABG).
* Have a condition that is likely to results in the episode of chest pain. The condition must be verified clinically during admission (i.e. pulmonary embolism, pneumonia, dissection of the aorta, …).
* Inflammatory joint disease.
* Insulin dependent diabetes.
* Fibromyalgia.
* Malignant disease.
* Apoplexy, dementia, or unable to cooperate.
* Major osseous anomaly.
* Osteoporosis.
* Pregnancy.
* Does not want to participate.
* Other - the reason for non-inclusion will be registered.

Exclusion Criteria:

Participants will be excluded following baseline evaluation if any of the following conditions are present

* Pain not related to the joints and muscles of the neck and/or thorax (CTA negative, see below).
* New incidence of any of the above mentioned conditions/pathologies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Worst chest pain during the last week. | 7 days
Patient-rated outcomes regarding improvement in chest pain. | 4 weeks

SECONDARY OUTCOMES:
Pain assessment | 7 days
Patient-specific disability (Patient Specific Functional Scale) | 4 weeks
SF-36 | 4 weeks
Global assessment(Improvement in chest pain and general health is rated by the participants using a 7-point scale) | 4 weeks
Direct health care cost, direct non-health care costs and indirect costs are used in as the economic indicator of cost-effectiveness. | 12 weeks
EQ-5D (modified version) | 4 weeks
Non-prescription medication use, visits to non-study health care providers, and time off work. | 12 weeks
Adverse events (Information about adverse events and side effects will be collected by the treating chiropractor after each treatment session.) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mette J Stochkendahl, DC, MSci, Principal Investigator — Nordic Institute of Chiropractic and Clinical Biomechanics; Jan Hartvigsen, DC, PhD, Study Chair — Nordic Institute of Chiropractic and Clinical Biomechanics and University of Southern Denmark
Locations (1):
- Dept. of Cardiology and Dept. of Nuclear Medicine, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Bechgaard P. [Segmentally thoracic pain in patients admitted to a coronary care unit]. Ugeskr Laeger. 1982 Jan 4;144(1):13-5. No abstract available. Danish. PMID 7064236
- [Background] Fruergaard P, Launbjerg J, Falch JF, Elsborg L, Hesse B, Jorgensen FB, Petri A, Mellemgaard K. [Differential diagnosis in acute chest pain and suspected myocardial infarction. A pilot study]. Ugeskr Laeger. 1992 Jan 13;154(3):138-41. Danish. PMID 1738954
- [Background] Capewell S, McMurray J. "Chest pain-please admit": is there an alternative?. A rapid cardiological assessment service may prevent unnecessary admissions. BMJ. 2000 Apr 8;320(7240):951-2. doi: 10.1136/bmj.320.7240.951. No abstract available. PMID 10753127
- [Background] Knockaert DC, Buntinx F, Stoens N, Bruyninckx R, Delooz H. Chest pain in the emergency department: the broad spectrum of causes. Eur J Emerg Med. 2002 Mar;9(1):25-30. doi: 10.1097/00063110-200203000-00007. PMID 11989492
- [Background] Spalding L, Reay E, Kelly C. Cause and outcome of atypical chest pain in patients admitted to hospital. J R Soc Med. 2003 Mar;96(3):122-5. doi: 10.1258/jrsm.96.3.122. PMID 12612112
- [Background] Fruergaard P, Launbjerg J, Hesse B, Jorgensen F, Petri A, Eiken P, Aggestrup S, Elsborg L, Mellemgaard K. The diagnoses of patients admitted with acute chest pain but without myocardial infarction. Eur Heart J. 1996 Jul;17(7):1028-34. doi: 10.1093/oxfordjournals.eurheartj.a014998. PMID 8809520
- [Background] Berman DS, Germano G, Shaw LJ. The role of nuclear cardiology in clinical decision making. Semin Nucl Med. 1999 Oct;29(4):280-97. doi: 10.1016/s0001-2998(99)80017-8. PMID 10534232
- [Background] Klocke FJ, Baird MG, Lorell BH, Bateman TM, Messer JV, Berman DS, O'Gara PT, Carabello BA, Russell RO Jr, Cerqueira MD, St John Sutton MG, DeMaria AN, Udelson JE, Kennedy JW, Verani MS, Williams KA, Antman EM, Smith SC Jr, Alpert JS, Gregoratos G, Anderson JL, Hiratzka LF, Faxon DP, Hunt SA, Fuster V, Jacobs AK, Gibbons RJ, Russell RO; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American Society for Nuclear Cardiology. ACC/AHA/ASNC guidelines for the clinical use of cardiac radionuclide imaging--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASNC Committee to Revise the 1995 Guidelines for the Clinical Use of Cardiac Radionuclide Imaging). Circulation. 2003 Sep 16;108(11):1404-18. doi: 10.1161/01.CIR.0000080946.42225.4D. No abstract available. PMID 12975245
- [Background] Launbjerg J, Fruergaard P, Hesse B, Jorgensen F, Elsborg L, Petri A. [The long-term prognosis of patients with acute chest pain of various origins]. Ugeskr Laeger. 1997 Jan 6;159(2):175-9. Danish. PMID 9012090
- [Background] Ockene IS, Shay MJ, Alpert JS, Weiner BH, Dalen JE. Unexplained chest pain in patients with normal coronary arteriograms: a follow-up study of functional status. N Engl J Med. 1980 Nov 27;303(22):1249-52. doi: 10.1056/NEJM198011273032201. PMID 7421961
- [Background] Eslick GD, Coulshed DS. Rapid assessment of chest pain. Chest pain clinics may be one step forward, two steps back. BMJ. 2002 Feb 16;324(7334):422. No abstract available. PMID 11855389
- [Background] Tew R, Guthrie EA, Creed FH, Cotter L, Kisely S, Tomenson B. A long-term follow-up study of patients with ischaemic heart disease versus patients with nonspecific chest pain. J Psychosom Res. 1995 Nov;39(8):977-85. doi: 10.1016/0022-3999(95)00065-8. PMID 8926607
- [Background] Wielgosz AT, Fletcher RH, McCants CB, McKinnis RA, Haney TL, Williams RB. Unimproved chest pain in patients with minimal or no coronary disease: a behavioral phenomenon. Am Heart J. 1984 Jul;108(1):67-72. doi: 10.1016/0002-8703(84)90546-5. PMID 6731285
- [Background] Achem SR, DeVault KR. Recent developments in chest pain of undetermined origin. Curr Gastroenterol Rep. 2000 Jun;2(3):201-9. doi: 10.1007/s11894-000-0062-4. PMID 10957931
- [Background] Christensen HW, Vach W, Gichangi A, Manniche C, Haghfelt T, Hoilund-Carlsen PF. Manual therapy for patients with stable angina pectoris: a nonrandomized open prospective trial. J Manipulative Physiol Ther. 2005 Nov-Dec;28(9):654-61. doi: 10.1016/j.jmpt.2005.09.018. PMID 16326234
- [Result] Stochkendahl MJ, Christensen HW, Vach W, Hoilund-Carlsen PF, Haghfelt T, Hartvigsen J. Chiropractic treatment vs self-management in patients with acute chest pain: a randomized controlled trial of patients without acute coronary syndrome. J Manipulative Physiol Ther. 2012 Jan;35(1):7-17. doi: 10.1016/j.jmpt.2010.11.004. Epub 2011 Dec 19. PMID 22185955
- [Result] Stochkendahl MJ, Christensen HW, Vach W, Hoilund-Carlsen PF, Haghfelt T, Hartvigsen J. A randomized clinical trial of chiropractic treatment and self-management in patients with acute musculoskeletal chest pain: 1-year follow-up. J Manipulative Physiol Ther. 2012 May;35(4):254-62. doi: 10.1016/j.jmpt.2012.04.003. PMID 22632585
- [Derived] Stochkendahl MJ, Sorensen J, Vach W, Christensen HW, Hoilund-Carlsen PF, Hartvigsen J. Cost-effectiveness of chiropractic care versus self-management in patients with musculoskeletal chest pain. Open Heart. 2016 May 4;3(1):e000334. doi: 10.1136/openhrt-2015-000334. eCollection 2016. PMID 27175285
- [Derived] Stochkendahl MJ, Christensen HW, Vach W, Hoilund-Carlsen PF, Haghfelt T, Hartvigsen J. Diagnosis and treatment of musculoskeletal chest pain: design of a multi-purpose trial. BMC Musculoskelet Disord. 2008 Mar 31;9:40. doi: 10.1186/1471-2474-9-40. PMID 18377636
- See also: Related Info — http://nikkb.dk